CLINICAL TRIAL: NCT03030703
Title: Salivary Cystatin SN Binds to Phytic Acid and is a Predictor of Non-heme Iron Bioavailability With Phytic Acid Supplementation
Brief Title: Cystatin SN Binds to Phytic Acid and Predicts Non-heme Iron Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: United States Department of Agriculture Foreign Agricultural Service (Other); American Academy of Nurse Practitioners (Unknown)
Responsible Party: Principal Investigator, Brian Lindshield, Ph.D., Associate Professor, Kansas State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SPPhyticAcidTrial
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia
Keywords: Phytic acid; Cystatin; Salivary proline-rich protein; antinutrient
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Phytic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 350 mg phytic acid (Experimental): 350 mg phytic acid (inositol hexaphosphate) at week 0 (before supplementation) and at week 4 (after supplementation)
  Interventions: Dietary Supplement: phytic acid

INTERVENTIONS:
Dietary Supplement: phytic acid — 350 mg phytic acid (inositol hexaphosphate) three times daily for four weeks
  Other Names: inositol hexaphosphate

SUMMARY:
Phytic acid is a known inhibitor of iron bioavailability, although long term studies have suggested possibly exaggerated findings compared to single meal studies, pointing to phytic acid adaptation over time. Salivary proline-rich proteins have been found to reduce tannin-iron chelation, but studies have not explored changes in salivary proteins that may result in phytic acid adaptation. The primary objectives of this study are: 1) To determine whether phytic acid impacts iron bioavailability or status when consumed over time 2) to test whether salivary protein production may impact iron bioavailability with phytic acid supplementation, and 3) to explore in vitro phytic acid salivary binding. Secondary objectives included assessment of the reliability of astringency as a measure of salivary protein production and iron absorption.

The study was conducted in an iron absorption study of 7 women, aged 18-35 years old, to determine iron bioavailability with supplementation of 350 mg phytic acid before and after regular, three times daily supplementation for four weeks. Direct iron absorption was measured using area under the curve. Iron status was measured by changes in hemoglobin and ferritin, and was adjusted by participant c-reactive protein levels. Salivary samples were collected before and after supplement consumption during meal challenges, and analyzed on HPLC and by ELISA. Astringency testing was conducted at the end of each meal challenge. In vitro saliva-phytic acid modeling was explored on HPLC, MALDI-TOF, and ELISA. Iron absorption and status markers were analyzed by ANOVA, and mixed-modeling followed by pairwise comparison by least significant differences. Pearson's correlations were used to correlated salivary proteins and astringency with iron bioavailability.

The present study will provide important information regarding the approximate influence of phytic acid consumption on iron bioavailability and storage over time in regards to salivary proteins. It will also give context to the role of salivary proteins with phytic acid consumption over time. Data will also help to delineate possible physiological mechanisms underlying phytic acid adaptation and possible ways to detect individuals who better adapt than others.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18-35 years' old
* Non-obese BMI (18-29.9)
* Signed informed consent

Exclusion Criteria:

* Oral disease
* Gastrointestinal disease
* Tobacco user
* Heavy alcohol user
* Pregnancy (assessed by pregnancy test)
* Lactation
* Medications affecting iron bioavailability
* Vitamin or mineral supplementation (other than vitamin B12)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Change in baseline to endline area under the curve after meal challenge at weeks 0 and 4 of intervention | Baseline and 4 weeks
  Change in area under the curve will be measured after administration of test meal including ferrous sulfate and condensed tannin supplementation at weeks 0 and 4
Change in baseline to endline hemoglobin and serum ferritin at weeks 0 and 4 of intervention | Baseline and 4 weeks
  Change in ferritin and hemoglobin will be measured before administration of test meals at weeks 0 and 4
Change in salivary proteins at weeks 0 and 4 of intervention | Baseline and 4 weeks
  HPLC determination of salivary proteins will be analyzed from saliva collected before and after test meals at weeks 0 and 4 of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Lindshield, Ph.D., Principal Investigator — Kansas State University
Locations (1):
- Physical Activity and Nutrition Research Consortium, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No